CLINICAL TRIAL: NCT06986811
Title: First-in-paediatrics, Open Label, Exploratory, Externally Controlled Clinical Trial to Evaluate Safety, Efficacy and Pharmacokinetics of 7-ethyl-10-hydroxy Camptothecin (SN-38) Formulated as a Biocompatible Polymeric Nanofiber Membrane (CEB-01) for Treatment, in Addition to Standard of Care, of Paediatric Patients From Birth to Less Than 18 Years of Age With a Locally Resectable Tumours in Comparison to Standard of Care
Brief Title: CEB-01 in Paediatrics With Locally Resectable Abdominal Tumours
Acronym: CEB-01-RLP01-C
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CEBIOTEX (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEB-01-RLP01-CT; 2024-520054-38-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Locally Resectable Paediatric Tumours
Keywords: CEB-01; SN-38; Locally resectable paediatrics tumours

STUDY DESIGN:
Intervention Model Description: 60 participants, open label treatment arm CEB-01 plus standard of care (consisting of surgery with/without radiotherapy and/or chemotherapy), compared with a well-matched population of approximately 10 patients, from the same participating sites, including historical controls (e.g. within the last 10 years) or contemporary controls (e.g. subjects that fulfil inclusion and exclusion criteria, but do not desire to receive experimental treatment) treated with standard of care (consisting of surgery with/without radiotherapy and/or chemotherapy) will be the external control arm.
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a single-blind trial in which investigators, and investigators' staff, will be aware of the treatment allocation (CEB-01 or not, but only once the tumour/ s removal has/have been completed). The participants, medical staff of the sponsor or data analysts will remain blinded to each participant's assigned study treatment from the time of randomization until database lock.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard surgery and CEB-01 implant after surgery (Experimental): Procedure/Surgery: Standard surgery The location and size of the tumor determine the type of surgery. Drug: CEB-01 It is novel formulation for local release of chemotherapy. It consists of a biocompatible and biodegradable nanofiber membrane made of poly(lactic-co-glycolic acid) (PLGA), which is loaded with the anti-tumor drug SN-38 and implanted in the surgical bed after tumor removal.
  Interventions: Procedure: Standard surgery; Drug: CEB-01
- Active Comparator: Arm 2 standard surgery (Active Comparator): Procedure/Surgery: Standard surgery The location and size of the tumor determine the type of surgery.
  Interventions: Procedure: Standard surgery

INTERVENTIONS:
Procedure: Standard surgery — The location and size of the tumor determine the type of surgery.
Drug: CEB-01 — It is novel formulation for local release of chemotherapy. It consists of a biocompatible and biodegradable nanofiber membrane made of poly(lactic-co-glycolic acid) (PLGA), which is loaded with the anti-tumor drug SN-38 and implanted in the surgical bed after tumor removal.
  Arms: Standard surgery and CEB-01 implant after surgery

SUMMARY:
The CEB-01 implant is a membrane containing SN-38, the active metabolite of irinotecan, an already authorized chemotherapeutic agent. After surgical removal of the abdominal cancer tumor, CEB-01 will be placed in the surgical bed for a local and sustained release of the chemotherapy. This is expected to delay or prevent local recurrence of abdominal tumors after surgery, while keeping a tolerable toxicity profile.

The study aims to assess the safety, tolerability, pharmacokinetics, and efficacy of CEB-01 in pediatric patients with locally resectable abdominal tumors including Soft Tissue Sarcoma (STS), high-risk Neuroblastoma (NB), Wilms tumour (WT), germ cell tumors (GCT), extracranial malignant rhabdoid tumour (eMRT), synovial sarcoma (SS), desmoplastic small round cell tumour (DSRCT) and fibrolamellar hepatocellular carcinoma (FL-HCC

DETAILED DESCRIPTION:
CEB-01-RLP01-CT trial is first-in-paediatrics, open label, exploratory, externally controlled clinical trial to evaluate safety, efficacy and pharmacokinetics of 7-ethyl-10-hydroxy-camptothecin (SN-38) formulated as a biocompatible polymeric nanofiber membrane (CEB-01) for treatment, in addition to standard of care, of paediatric patients from birth to less than 18 years of age with de novo or recurrent, locally resectable, abdominal tumors in comparison to standard of care.

The trial population will consist of 80 participants who fulfil all the inclusion and exclusion criteria, allocated in three cohorts:

Cohort 1: 20 participants with abdominal STS, open label treatment arm consisting of CEB-01 plus the standard of care (which may include surgery, with or without radiotherapy and/or chemotherapy). The outcomes will be compared to a well-matched population of about 10 participants from the same participating sites, including historical controls or contemporary controls.

Cohort 2: 20 participants with high-risk NB, open label treatment arm consisting of CEB-01 plus the standard of care (which may include surgery, with or without radiotherapy and/or chemotherapy). The outcomes will be compared to a well-matched population of about 10 participants from the same participating sites, including historical controls or contemporary controls.

Cohort 3: 20 participants with rare abdominal tumors including WT, GCT, eMRT, SS, DSRCT and FL-HCC, open label uncontrolled treatment arm to obtain additional safety and efficacy data.

For measurement of primary safety and efficacy endpoints, follow-up will consist of short-term evaluation at 365 ± 30 days and long-term evaluation at 1095 ± 30 days post-surgery as it is considered sufficient for the assessment of the therapeutic effect of CEB-01 regarding local recurrence.

For pharmacokinetic assessment, blood samples will be collected at baseline and at 9 different time points until 56 ± 7 days post-surgery.

For each participant the trial duration will be composed of a screening period for up to 28 days, one day for surgery and 1095 ± 30 days of follow-up.

A Data Safety Monitoring Board (DSMB) will review data in an unblinded fashion; details are given in the DSMB charter. ScheduledThe scheduled review will be performed by the DSMB once 10 randomised and treated participants have completed 6 months of follow-up. The DSMB can be convened at the request of the sponsor should safety signals be detected

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this trial, an individual must meet all the following criteria:

1. ≤ 18 years.
2. Participants must have a diagnosis of:

   1. De novo or recurrent abdominal soft-tissue sarcoma.
   2. De novo or recurrent high-risk neuroblastoma according to Children's Oncology Group (COG) risk classification, regardless of response to frontline therapy, diagnosed either by a former histologic verification of neuroblastoma and/or former demonstration of tumour cells in the bone marrow with increased urinary catecholamines at the time of study enrolment. Participants who were initially considered low or intermediate risk but were then reclassified as high risk are also eligible.
   3. Other tumours: recurrent Wilms tumour, de novo or recurrent Germ cell tumour, de novo or recurrent extracranial malignant rhabdoid tumour, de novo or recurrent synovial sarcoma, de novo or recurrent fibrolamellar hepatocellular carcinoma, and de novo or recurrent desmoplastic small round cell tumour.
3. A histology assessment is required for enrolment of de novo cases. A new histology assessment is not required for enrolment of the recurrent cases, but it will be obtained from the resected tumour to assess whether the histology is identical to the original tumour.
4. Participants previously treated with irinotecan will be eligible if they have not had documented progressive disease during treatment.
5. Participants might have more than one surgically removable lesion.
6. Adequate liver, renal, haematological, and cardiac function.
7. Participants must have fully recovered from the acute toxic effects (Grade 3 or above) of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this trial.
8. Landky or Karnosfsky functional performance status score ≥ 50 at screening.
9. Female participants of childbearing potential must have a negative urine betahuman chorionic gonadotropin (beta-hCG) pregnancy test at time of screening.
10. Female and male participants of childbearing potential must be willing to use adequate contraception throughout the study and for 6 months after surgery.
11. Life expectancy greater than 6 months.
12. The participant legally authorized guardian must acknowledge in writing that consent to become a study subject has been obtained prior to any protocol screening procedures.

Exclusion Criteria

An individual who meets any of the following criteria will be excluded from participation in this trial:

1. Metastatic lesions.
2. Other malignancies within past 2 years except for in-situ cancers or basal/squamous cell skin cancer. Subjects with other malignancies are eligible if they are disease-free for at least 24 months or have a clinically stable concurrent malignancy not requiring tumour-directed treatment.
3. Active bacterial, viral or fungal infection.
4. Known history of active human immunodeficiency virus (HIV) infection, hepatitis B, hepatitis C or chronic liver disease. Testing is not required in the absence of clinical findings or suspicion.
5. Impossibility of ensuring adequate follow-up.
6. Participants who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.
7. Contraindication to computed tomography (CT) scan.
8. Major surgery within 14 days prior to the implant of study drug or still in recovery after experiencing surgical complications; neither tumour biopsy nor central line insertion are considered a major surgery.
9. Other relevant concomitant illnesses.
10. Participant' status post-allogeneic stem cell transplant are not eligible.
11. Participants with disease of any major organ system that would compromise their ability to withstand therapy.
12. Patients with tumour size requiring CEB-01 implant that exceeds the maximum implantable surface area based on Body Surface Area (BSA) correction.
13. Patients with known hypersensitivity to SN-38 or any of the CEB-01 excipients.
14. Pregnancy or lactation. Pregnant women are excluded from this study; if the patient is a lactating mother, breastfeeding should be discontinued.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Frequency of Adverse Events (AEs) (Safety) | Through study completion, average 3 years
  Adverse Events (AE), serious and non-serious, with their frequency, severity, and relatedness to study drug and coded according to the most updated version of the Common Terminology Criteria for Adverse Events (CTCAE).

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Through study completion, average 3 years
  Defined as the time from surgery to objective tumour progression or death from any cause.
Overall survival (OS). | Through study completion, average 3 years
  Defined as time from surgery to death from any cause.
Local recurrence-free survival (LRFS) | Through study completion, average 3 years
  Defined as the time from surgery until the progression of the disease in the area of implanted CEB-01.
New lesions either distant or metastatic by RECIST 1.1 (Response Evaluation Criteria in Solid Tumors, version 1.1) | Through study completion, average 3 years
  Number of new lesions either distant or metastatic by RECIST 1.1. (Response Evaluation Criteria in Solid Tumors, version 1.1)
Area under the concentration-time curve (AUC0-inf) of SN-38 ( 7-ethyl-10-hydroxy Camptothecin) | During 60 days
  Represents the total SN-38 (f 7-ethyl-10-hydroxy Camptothecin) exposure in the peripheral blood across time
Maximum concentration (Cmax) of SN-38. | During 60 days
  The highest concentration of SN-38 in the peripheral blood samples taken at sequential timepoints
Time of maximum plasma concentration (Tmax) of SN38. | During 60 days
  Time from the surgery to the moment with the highest concentration of SN-38 in the peripheral blood samples taken at sequential timepoints
Terminal half-life (t1/2) of SN-38 | During 60 days
  he time required for the plasma concentration of SN-38 to fall by 50% from the Cmax

CONTACTS AND LOCATIONS:
Overall Officials: Marta Pilar Martin Gimenez, M.D.; Ph.D., Principal Investigator — Hospital Sant Joan de Deu
Locations (1):
- Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be provided.